CLINICAL TRIAL: NCT01017601
Title: A Randomized Double-Blinded Phase II Study of NTX-010, a Replication-Competent Picornavirus, After Standard Platinum-Containing Cytoreductive Induction Chemotherapy in Patients With Extensive Stage Small Cell Lung Cancer
Brief Title: Seneca Valley Virus-001 After Chemotherapy in Treating Patients With Extensive-Stage Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Interim analysis declared futility.
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCCTG-N0923; NCCTG-N0923; CDR0000659547 (Registry Identifier: PDQ (Physician Data Query)); NCI-2011-01991 (Registry Identifier: CTRP (Clinical Trials Reporting System))
Record Dates: First submitted 2009-11-19; First posted 2009-11-20 (Estimated); Results first posted 2017-05-08 (Actual); Last update posted 2017-05-08 (Actual); Status verified 2017-03

CONDITIONS: Lung Cancer
Keywords: extensive stage small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients receive a single dose of Seneca Valley virus-001 (NTX-010) IV over 1 hour on day 1.
  Interventions: Biological: Seneca Valley virus-001
- Arm II (Placebo Comparator): Patients receive a single dose of placebo IV over 1 hour on day 1.
  Interventions: Other: placebo

INTERVENTIONS:
Biological: Seneca Valley virus-001 — Given IV
  Arms: Arm I
Other: placebo — Given IV
  Arms: Arm II

SUMMARY:
RATIONALE: A virus called Seneca Valley virus-001 (NTX-010) may be able to kill tumor cells without damaging normal cells. It is not yet known whether NTX-010 is more effective than a placebo in treating small cell lung cancer.

PURPOSE: This randomized phase II trial is studying NTX-010 to see how well it works compared with a placebo when given after chemotherapy in treating patients with extensive-stage small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare the progression-free survival (PFS) of patients with extensive-stage small cell lung cancer treated with Seneca Valley virus-001 (NTX-010) vs placebo.

Secondary

* To compare the overall survival (OS) of patients treated with NTX-010 vs placebo.
* To describe the adverse events profile and safety of NTX-010 in this patient population.
* To determine the antitumor response rate, as assessed by RECIST criteria, and duration of tumor response in this patient population.
* To assess the quality of life of this patient population.

Exploratory

* To determine the relationship between the presence of neutralizing antibodies and PFS.
* To assess whether or not a slow viral clearance is associated with better response as determined by PFS.
* To determine any potential impact of the presence of one or several neuroendocrine markers in the tumor sample (synaptophysin, chromogranin, or CD56) on PFS and OS.
* To determine any potential relationship between presence of cell surface determinants of NTX-010 tropism in the tumor tissue and clinical outcomes such as improved PFS and OS.
* To determine any potential relationship between the loss of integrity of IFN signaling in the tumor tissue and clinical outcomes such as improved PFS and OS.
* To assess whether or not the presence of circulating tumor cells permissive to NTX-010 is associated with better clinical outcomes as determined by PFS and OS.

OUTLINE: This is a multicenter study. Patients are stratified according to ECOG performance status (0 vs 1), tumor response to standard chemotherapy (partial response vs stable disease vs complete response), and time between completion of chemotherapy to randomization 1 month (≤1 month) vs 2 months (>1 month but ≤ 2 months) vs 3 months (> 2 months but ≤ 3 months). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive a single dose of Seneca Valley virus-001 (NTX-010) IV over 1 hour on day 1.
* Arm II: Patients receive a single dose of placebo IV over 1 hour on day 1. In both arms, patients may also undergo prophylactic cranial irradiation (PCI) daily on days 22-35 if they have not previously undergone PCI or whole-brain radiotherapy.

Quality of life is assessed at baseline and then periodically during the study.

Blood samples are collected periodically for viral clearance and antiviral neutralizing antibody levels, circulating tumor cells, and other biomarker laboratory studies.

After completion of study therapy, patients are followed up periodically for up to 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of extensive-stage small cell lung cancer (SCLC)

  * No mixed histology
* Presence of ≥ 1 neuroendocrine marker (synaptophysin, chromogranin, or CD56) in tumor tissue
* Achieved partial response (PR), complete response (CR), or stable disease (SD) ≤ 12 weeks of completing 4-6 courses of platinum-based chemotherapy regimen for extensive-stage SCLC

  * Patients with PR or SD must have measurable disease, defined as ≥ 1 lesion whose longest diameter can be accurately measured as ≥ 2.0 cm but < 10 cm by chest x-ray OR as ≥ 1.0 cm but < 10 cm by CT scan, CT component of a PET/CT scan, or MRI

    * If CT scan is used, it must be used for both pre- and post-treatment tumor assessments
    * Measurable disease is not required for patients with CR
* Brain metastases allowed provided they have been stable for ≥ 4 weeks after completion of prior radiotherapy

PATIENT CHARACTERISTICS:

* ECOG performance status 0 or 1
* Life expectancy of ≥ 8 weeks
* ANC ≥ 1,500/μL
* Platelet count ≥ 100,000/μL
* Hemoglobin ≥ 9 g/dL
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN) OR direct bilirubin normal
* AST ≤ 3 times ULN (≤ 5 times ULN if liver has tumor involvement)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use adequate contraception
* Able to comply with study procedures to minimize virus exposure to others
* Willing to provide required biologic specimens
* Willing to return to NCCTG/CTSU enrolling institution for follow-up
* Adequate lung function (i.e., not oxygen dependent)

  * The patient is eligible if not on a 24-hour oxygen schedule
* No second primary malignancy within the past 5 years, except for the following:

  * Carcinoma in situ of the cervix
  * Non-melanomatous skin cancer
  * History of low-grade (Gleason score ≤ 6) localized prostate cancer (even if diagnosed < 5 years prior to study entry)
  * Stage I breast cancer that was treated ≥ 5 years before study entry
  * Transitional cell carcinoma of the bladder (in situ)
* No active hepatitis B or hepatitis C
* No clinically significant infection
* No significant traumatic injury within the past 4 weeks
* No concurrent uncontrolled illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situation that would limit compliance with study requirements

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 4 weeks since prior radiotherapy (2 weeks for palliative radiotherapy to skeletal metastases)
* Other prior radiation therapy (including WBRT, PCI, or Gamma Knife) is permitted as long as the following are true:

  * Recovered from prior radiotherapy (alopecia allowed)
  * No prior consolidation radiation therapy to the chest
  * No prior radiotherapy to > 25% of bone marrow
  * For patients without brain metastases, WBRT or standard of care PCI completed ≥ 2 weeks before administration of NTX- 010/placebo
* More than 365 days since prior immunotherapy or biologic therapy
* More than 4 weeks since prior major surgery* (i.e., laparotomy) or open biopsy
* More than 2 weeks since prior minor surgery*
* No prior exposure to the Seneca Valley virus (NTX-010), as determined by negative serum antibodies
* No concurrent combination antiretroviral therapy for HIV-positive patients NOTE: *Insertion of a vascular access device is not considered major or minor surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2010-01; Primary Completion 2013-01 (Actual); Study Completion 2014-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julian Molina, MD, PhD, Study Chair — Mayo Clinic
Locations (196):
- United States (196):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Valley Medical Oncology Consultants - Castro Valley, Castro Valley, California
  - Valley Medical Oncology, Fremont, California
  - Contra Costa Regional Medical Center, Martinez, California
  - El Camino Hospital Cancer Center, Mountain View, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Breast Surgeons, Incorporated, Oakland, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Larry G Strieff MD Medical Corporation, Oakland, California
  - Tom K Lee, Incorporated, Oakland, California
  - Epic Care - Oakland, Oakland, California
  - Doctors Medical Center - San Pablo Campus, San Pablo, California
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - George Bray Cancer Center at the Hospital of Central Connecticut - New Britain Campus, New Britain, Connecticut
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Saint Alphonsus Cancer Care Center at Saint Alphonsus Regional Medical Center, Boise, Idaho
  - St. Joseph Regional Medical Center, Lewiston, Idaho
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Elkhart Clinic, LLC, Elkhart, Indiana
  - Michiana Hematology-Oncology, PC - Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Michiana Hematology-Oncology, PC - South Bend, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center, Mishawaka, Indiana
  - Michiana Hematology Oncology PC - Plymouth, Plymouth, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC - La Porte, Westville, Indiana
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, Clive, Iowa
  - Mercy Cancer Center - West Lakes, Clive, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Liberal, Liberal, Kansas
  - Cancer Center of Kansas, PA - McPherson, McPherson, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Ochsner Cancer Institute at Ochsner Clinic Foundation, New Orleans, Louisiana
  - York Hospital's Oncology Treatment Center, York Village, Maine
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Lakeside Cancer Specialists, PLLC, Saint Joseph, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - MeritCare Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology - Woodbury, Woodbury, Minnesota
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Roswell Park Cancer Institute, Buffalo, New York
  - Tucker Center for Cancer Care at Orange Regional Medical Center, Middletown, New York
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - FirstHealth Moore Regional Community Hospital Comprehensive Cancer Center, Pinehurst, North Carolina
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - Roger Maris Cancer Center at MeritCare Hospital, Fargo, North Dakota
  - Wood County Oncology Center, Bowling Green, Ohio
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Community Cancer Center, Elyria, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - UPMC Cancer Centers, Pittsburgh, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Erlanger Cancer Center at Erlanger Hospital - Baroness, Chattanooga, Tennessee
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Overlake Cancer Center at Overlake Hospital Medical Center, Bellevue, Washington
  - Providence Centralia Hospital, Centralia, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - St. Francis Hospital, Federal Way, Washington
  - Providence St. Peter Hospital Regional Cancer Center, Olympia, Washington
  - Good Samaritan Cancer Center, Puyallup, Washington
  - Rockwood Clinic Cancer Treatment Center, Spokane, Washington
  - Franciscan Cancer Center at St. Joseph Medical Center, Tacoma, Washington
  - Allenmore Hospital, Tacoma, Washington
  - CCOP - Northwest, Tacoma, Washington
  - MultiCare Regional Cancer Center at Tacoma General Hospital, Tacoma, Washington
  - St. Clare Hospital, Tacoma, Washington
  - Marshfield Clinic Cancer Care at Regional Cancer Center, Eau Claire, Wisconsin
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Holy Family Memorial Medical Center Cancer Care Center, Manitowoc, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Marshfield Clinic - Lakeland Center, Minocqua, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Ministry Medical Group at Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin
  - St. Nicholas Hospital, Sheboygan, Wisconsin
  - Marshfield Clinic at Saint Michael's Hospital, Stevens Point, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

REFERENCES:
- [Derived] Schenk EL, Mandrekar SJ, Dy GK, Aubry MC, Tan AD, Dakhil SR, Sachs BA, Nieva JJ, Bertino E, Lee Hann C, Schild SE, Wadsworth TW, Adjei AA, Molina JR. A Randomized Double-Blind Phase II Study of the Seneca Valley Virus (NTX-010) versus Placebo for Patients with Extensive-Stage SCLC (ES SCLC) Who Were Stable or Responding after at Least Four Cycles of Platinum-Based Chemotherapy: North Central Cancer Treatment Group (Alliance) N0923 Study. J Thorac Oncol. 2020 Jan;15(1):110-119. doi: 10.1016/j.jtho.2019.09.083. Epub 2019 Oct 9. PMID 31605793

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One-hundred twenty-one (121) participants were pre-registered and 59 participants were registered between January 2010 and January 2013. Study was terminated prematurely on 1/10/2013 due to an interim analysis that declared futility. No additional clinical and survival follow-up data are required as of 11/15/2014.
Pre-assignment Details: Sixty-two participants were deemed screen failures: 26 progression, 21 did not meet eligibility criteria, 6 patient decision and 9 other reason. Out of the 59 randomized participants, there were 8 cancellations and one participant was found to be ineligible upon audit. All seventy-one participants mentioned above were excluded from all analyses.
Groups:
- Arm I (NTX-010): Patients receive a single dose of Seneca Valley virus-001 (NTX-010) IV over 1 hour on day 1.
- Arm II (Placebo): Patients receive a single dose of placebo IV over 1 hour on day 1.
Period: Overall Study
Arm/Group | Arm I (NTX-010) | Arm II (Placebo)
Started | 26 | 24
Completed | 14 | 11
Not Completed | 12 | 13
Not completed — Disease Progression | 12 | 12
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: All registered participants who have met eligibility criteria and started the treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (NTX-010) | Arm II (Placebo) | Total
Number analyzed (Participants) | 26 | 24 | 50
Age, Continuous [Median (Full Range); unit: years] | 67 [44 to 81] | 60 [50 to 82] | 63 [44 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 26
  Male | 14 | 10 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 24 | 24 | 48
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 26 | 24 | 50
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants]
  0=Asymptomatic and fully active | 8 | 7 | 15
  1=Symptomatic and fully ambulatory | 18 | 17 | 35
Prior Response to Chemo [Count of Participants; unit: Participants]
  Stable Disease (SD) | 4 | 5 | 9
  Partial Response (PR) | 15 | 12 | 27
  Complete Response (CR) | 7 | 7 | 14
Cigarette History [Count of Participants; unit: Participants]
  Never Smoked | 0 | 2 | 2
  Current Smoker | 7 | 4 | 11
  Former Smoker | 19 | 18 | 37
Time between Completion of Chemo to Randomization [Count of Participants; unit: Participants]
  1 month | 10 | 9 | 19
  2 months | 10 | 10 | 20
  3 months | 6 | 4 | 10
  Unknown | 0 | 1 | 1
Prior Radiation Therapy [Count of Participants; unit: Participants]
  Yes | 8 | 9 | 17
  No | 18 | 15 | 33
Enrolling Group [Count of Participants; unit: Participants]
  Previously untreated | 3 | 4 | 7
  Previously treated | 23 | 20 | 43

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: The progression-free survival (PFS) was defined as the time from date of randomization to the documentation of disease progression or death as a result of any cause, whichever comes first.
Time Frame: Time from randomization to the disease progression or death (up to 5 years)
Population: All registered participants who have met eligibility criteria and started the treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (NTX-010) | Arm II (Placebo)
Number analyzed (Participants) | 26 | 24
months | 1.7 [1.4 to 3.1] | 1.7 [1.4 to 4.3]

2. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from study enrollment (randomization) to the time of death from any cause or last follow-up.
Time Frame: Time from randomization to death or last follow-up (up to 5 years)
Population: All registered participants who have met eligibility criteria and started the treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (NTX-010) | Arm II (Placebo)
Number analyzed (Participants) | 26 | 24
months | 6.6 [4.7 to 13.2] | 13.1 [5.8 to 19.0]

3. Secondary Outcome: Response Rate (Complete Response and Partial Response) as Assessed by Response Evaluation Criteria in Solid Tumors (RECIST)
Description: A confirmed tumor response was defined as a complete response (CR) or partial response (PR) noted as the objective status on 2 consecutive evaluations at least 6 weeks apart. Response and progression will be evaluated in this study using the new international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1). Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all non-nodal target lesions and each target lymph node must have reduction in short axis to <1.0 cm.; Partial Response (PR), at least a 30% decrease in the sum of the longest diameters of the non-nodal target lesions and the short axes of the target lymph nodes taking as reference the Baseline Sum of Diameters; Overall Response (OR) = CR + PR.
Time Frame: Up to 5 years
Population: All registered participants who have met eligibility criteria and started the treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Arm I (NTX-010) | Arm II (Placebo)
Number analyzed (Participants) | 26 | 24
percentage of participants
  Confirmed Response (CR/PR) | 3.9 | 16.6
  Stable Disease (SD) | 15.4 | 8.3
  Progression Disease (PD) | 73.1 | 75.0
  Non-CR/non-PD | 3.9 | 0
  Not evaluable | 3.9 | 0

4. Secondary Outcome: Duration of Response
Description: Duration of response was defined as the time from the date at which the patient's earliest best objective status was first noted to be either a CR or PR to the earliest date progression was documented.
Time Frame: Up to 5 years
Population: All participants with the patient's earliest best objective status was first noted to be a CR or PR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (NTX-010) | Arm II (Placebo)
Number analyzed (Participants) | 4 | 4
months | 1.9 [1.4 to 19.4] | NA [3.2 to NA] — Two participants had disease progression. Median time and the upper limit of 95% CI are unattainable.

5. Secondary Outcome: Number of Participants With at Least One Grade 3 or Above Adverse Events Assessed by NCI CTCAE v4.0
Description: Adverse events were assessed by Common Terminology Criteria for Adverse Events (CTCAE) v4.0. Grading: Grade 1=Mild, Grade 2=Moderate, Grade 3=Severe, Grade 4=Life-threatening, Grade 5=Death. The maximum grade for each type of adverse events were recorded for each patient.
Time Frame: Up to 23 months
Population: All registered participants who have met eligibility criteria and started the treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (NTX-010) | Arm II (Placebo)
Number analyzed (Participants) | 26 | 24
Participants | 9 | 5

6. Secondary Outcome: Change From Baseline to Day 20-29 in the LASA QOL
Description: Quality of Life (QOL) was measured using the single-item Linear Analogue Self Assessment (LASA) on a 0-10 scale, with 0=as bad as it can be and 10=as good as it can be. The QOL scores was converted to a 100-point scale, with 0=Low QOL and 100=Best QOL. Change from baseline to day 20-29 was calculated by subtracting the baseline scores from the scores at day 20-29. Negative change indicates the QOL decrease and positive change indicates the QOL improvement.
Time Frame: Day 1 Cycle 1 prior to treatment (baseline) and day 20-29 (during the active monitoring phase)
Population: All registered participants who have met eligibility criteria and who have completed both baseline and the time point of day 20-29 QOL assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm I (NTX-010) | Arm II (Placebo)
Number analyzed (Participants) | 10 | 7
units on a scale | -9.0 (17.9) | -5.7 (31.0)
Statistical Analysis 1: Comparison: Arm I (NTX-010) vs Arm II (Placebo); Test type: Other; p = 0.50, Wilcoxon Rank Sum

7. Secondary Outcome: Change From Baseline to Day 30-59 in the LASA QOL
Description: Quality of Life (QOL) was measured using the single-item Linear Analogue Self Assessment (LASA) on a 0-10 scale, with 0=as bad as it can be and 10=as good as it can be. The QOL scores was converted to a 100-point scale, with 0=Low QOL and 100=Best QOL. Change from baseline to day 30-59 was calculated by subtracting the baseline scores from the scores at day 30-59. Negative change indicates the QOL decrease and positive change indicates the QOL improvement.
Time Frame: Day 1 Cycle 1 prior to treatment (baseline) and day 30-59 (during the active monitoring phase)
Population: All registered participants who have met eligibility criteria and who have completed both baseline and the time point of day 30-59 QOL assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm I (NTX-010) | Arm II (Placebo)
Number analyzed (Participants) | 9 | 10
units on a scale | -6.7 (26.0) | -1.0 (11.0)
Statistical Analysis 1: Comparison: Arm I (NTX-010) vs Arm II (Placebo); Test type: Other; p = 0.96, Wilcoxon Rank Sum

8. Secondary Outcome: Clinical Significance Change From Baseline to Day 20-29 in the LASA QOL
Description: Quality of Life (QOL) was measured using the single-item Linear Analogue Self Assessment (LASA) on a 0-10 scale, with 0=as bad as it can be and 10=as good as it can be. The QOL scores was converted to a 100-point scale, with 0=Low QOL and 100=Best QOL. Change from baseline to day 20-29 was calculated by subtracting the baseline scores from the scores at day 20-29. Clinical Significance change over time was determined by the percentage of patients that report an improvement of more than 10 points on the 0-100 point scale.
Time Frame: Day 1 Cycle 1 prior to treatment (baseline) and day 20-29 (during the active monitoring phase)
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Arm I (NTX-010) | Arm II (Placebo)
Number analyzed (Participants) | 10 | 7
percentage of participants | 10 | 28.6
Statistical Analysis 1: Comparison: Arm I (NTX-010) vs Arm II (Placebo); Test type: Other; p = 0.54, Fisher Exact

9. Secondary Outcome: Clinical Significance Change From Baseline to Day 30-59 in the LASA QOL
Description: Quality of Life (QOL) was measured using the single-item Linear Analogue Self Assessment (LASA) on a 0-10 scale, with 0=as bad as it can be and 10=as good as it can be. The QOL scores was converted to a 100-point scale, with 0=Low QOL and 100=Best QOL. Change from baseline to day 30-59 was calculated by subtracting the baseline scores from the scores at day 30-59. Clinical Significance change over time was determined by the percentage of patients that report an improvement of more than 10 points on the 0-100 point scale.
Time Frame: Day 1 Cycle 1 prior to treatment (baseline) and day 30-59 (during the active monitoring phase)
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Arm I (NTX-010) | Arm II (Placebo)
Number analyzed (Participants) | 9 | 10
percentage of participants | 22.2 | 20.0
Statistical Analysis 1: Comparison: Arm I (NTX-010) vs Arm II (Placebo); Test type: Other; p = 1.0, Fisher Exact

ADVERSE EVENTS:
Time Frame: Up to 23 months
Description: All registered participants who have met eligibility criteria and started the treatment.
Arm/Group | Arm I (NTX-010) | Arm II (Placebo)
Serious Adverse Events (participants affected / at risk) | 1/26 | 0/24
Other Adverse Events (participants affected / at risk) | 24/26 | 17/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (NTX-010) (N=26) | Arm II (Placebo) (N=24)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (NTX-010) (N=26) | Arm II (Placebo) (N=24)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 8 (11) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 8 (10) | 1 (1)
Flu like symptoms (General disorders) | 16 (20) | 6 (9)
Mucosal infection (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 1 (1)
Creatinine increased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (2) | 1 (1)
Weight loss (Investigations) | 5 (13) | 5 (15)
White blood cell decreased (Investigations) | 2 (2) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (4) | 1 (2)
Musculoskeletal deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Brachial plexopathy (Nervous system disorders) | 0 (0) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 1 (4) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (3) | 1 (5)
Confusion (Psychiatric disorders) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (10) | 9 (18)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less